CLINICAL TRIAL: NCT07124650
Title: Effect of Hydrocortisone and Lidocaine on Endotracheal Tube for Sore Throat and Hoarseness After Thyroid/Parathyroid Surgery With Neuromonitoring: A Randomized Controlled Trial
Brief Title: Sore Throat After Open Neck Elective Surgery
Acronym: STONES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Saint Petersburg State University, Russia (Other)
Collaborators: Smooth Drug Development (Unknown)
Responsible Party: Principal Investigator, Efremov Sergey, Deputy director for science, Saint-Petersburg state university hospital, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPbU-STONES-2025
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Sore Throat, Cough, Hoarseness; Thyroid and Parathyroid Surgery
Keywords: Hydrocortisone; Lidocaine; Endotracheal tube; Neuromonitoring; Randomized controlled trial
MeSH Terms: conditions — Cough; Hoarseness; Thyroid Diseases | interventions — hydrocortisone acetate; Ointments; Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydrocortisone group (Experimental): Participants receive endotracheal tubes coated with 1% hydrocortisone ointment to reduce postoperative sore throat and hoarseness.
  Interventions: Drug: Hydrocortisone Acetate 1% Ointment
- Lidocaine group (Experimental): Participants receive endotracheal tubes coated with 0.05% lidocaine and chlorhexidine solution (Cathelgel).
  Interventions: Drug: Lidocaine hydrochloride 0,05% with chlorhexidine

INTERVENTIONS:
Drug: Hydrocortisone Acetate 1% Ointment — Endotracheal tubes will be coated with 1% hydrocortisone acetate ointment prior to intubation. The ointment will be applied uniformly to the outer surface of the tube. This intervention aims to reduce postoperative throat inflammation and pain.
  Arms: Hydrocortisone group
Drug: Lidocaine hydrochloride 0,05% with chlorhexidine — Endotracheal tubes will be treated with 0.05% lidocaine hydrochloride solution combined with chlorhexidine (Cathejell). The solution will be applied to the tube surface before intubation to provide local anesthesia and reduce postoperative throat discomfort.
  Other Names: Cathejell
  Arms: Lidocaine group

SUMMARY:
This randomized, double-blind clinical trial aims to evaluate the effectiveness of two medications-hydrocortisone ointment and lidocaine solution-applied to the endotracheal tube in reducing postoperative throat pain, hoarseness, and cough following thyroid or parathyroid surgery with neuromonitoring.

A total of 764 adult patients undergoing elective neck surgery at Saint-Petersburg State University Hospital will be enrolled and randomly assigned to receive either a hydrocortisone-coated or lidocaine-coated endotracheal tube.

Outcomes will be assessed upon awakening from anesthesia, at 24 hours, and again at 3 days postoperatively.

The findings may contribute to improving postoperative comfort and recovery for patients undergoing similar surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective open surgery on the thyroid/parathyroid glands with intraoperative neuromonitoring.
* Age ≥18 years.
* Willing and able to provide voluntary informed consent for participation in the study.

Exclusion Criteria:

* Pregnancy (for women of childbearing potential).
* Known allergy to hydrocortisone or lidocaine.
* Refusal to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 764 (Estimated)
Dates: Start 2025-09-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Frequency of severe throat pain at 24 hours post-operation | 24 hours post-operation
  Proportion of patients scoring ≥3 points on the STONES throat pain subscale (0 = no pain, 1 = mild, 2 = moderate, 3 = severe pain) assessed 24 hours after thyroid/parathyroid surgery. Evaluated through patient-reported questionnaire administered by a blinded investigator.
Frequency of clinically significant EMG signal reduction | Perioperative/periprocedural
  Proportion of patients showing ≥50% decrease in amplitude of electromyographic (EMG) signals from recurrent laryngeal nerve during intraoperative neuromonitoring compared to baseline measurements (V1/ R1 timepoints), using the C2 neuromonitor system.

SECONDARY OUTCOMES:
Frequency of intraoperative laryngeal reflexes (coughing) | Perioperative/periprocedural
  Number of coughing episodes recorded by anesthesiologist during surgical procedure, graded as: 0 = no cough, 1 = single mild cough, 2 = persistent cough requiring intervention.
Episodes of complete EMG signal loss during surgery | Perioperative/periprocedural
  Number of events with total loss of electromyographic response (OmV amplitude) during stimulation of recurrent laryngeal nerve, confirmed by repeated measurements at standard timepoints (V1/R1 to V2/R2).
Vocal cord mobility impairment (laryngoscopy) | 72 hours after surgery
  Presence of unilateral/bilateral vocal cord paralysis or paresis detected through postoperative fiberoptic laryngoscopic examination, graded as: 0 = normal mobility, 1 = reduced mobility, 2 = complete paralysis."
Neck Disability Index (NDI) score | 3 days after surgery
  Patient-reported functional limitation score (0-50 scale) assessing neck pain impact on daily activities, with higher scores indicating greater disability. Collected through standardized questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey M. Efremov, MD, PhD, Principal Investigator — Saint Petersburg State University Hospital
Locations (1):
- Saint Petersburg State University Hospital, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Row data may be shared by the reasonable request
Supporting Information: Study Protocol, SAP